CLINICAL TRIAL: NCT00450112
Title: A Multi-Center Extension and Open-Label Study of a Single or Repeat Intra-Articular Injection of Gel-200 in Osteoarthritis of the Knee.
Brief Title: Gel-200 Extension and Open-Label Study in Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Responsible Party: Osamu Akahane, Seikagaku Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gel/1132
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Results first posted 2011-08-22 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-07

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Gel-200 — Single Intra-articular Injection

SUMMARY:
The purpose of this study is to determine if a single or repeat intra-articular injection of Gel-200 is safe and effective in subjects with symptomatic osteoarthritis of the knee and to determine if original SI-6606/01 Gel-200 therapy is durable beyond the original study.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in study SI-6606/01.

Exclusion Criteria:

* Female subjects who are pregnant or lactating.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SKK, Plantation, Florida, United States

REFERENCES:
- [Derived] Takamura J, Seo T, Strand V. A Pooled Analysis of Two Multicenter, Randomized Controlled Trials of a Single Intra-articular Injection of Gel-200 for Treatment of Osteoarthritis of the Knee. Clin Med Insights Arthritis Musculoskelet Disord. 2018 May 9;11:1179544118773068. doi: 10.1177/1179544118773068. eCollection 2018. PMID 29780263
- [Derived] Strand V, Lim S, Takamura J. Evidence for safety of retreatment with a single intra-articular injection of Gel-200 for treatment of osteoarthritis of the knee from the double-blind pivotal and open-label retreatment clinical trials. BMC Musculoskelet Disord. 2016 Jun 1;17:240. doi: 10.1186/s12891-016-1101-0. PMID 27250845

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 202 patients were entered.
Groups:
- 2Gel-200: Patients already received 1 single dose of Gel-200 (3 mL) and followed up for 13 weeks in previous study(NCT00449696). After completion of previous study, patients entered this study and received 1 single dose of Gel-200 (3mL) intra-articular injection again into knee joint.
- 1PBS1Gel-200: Patients already received 1 single dose of Phosphate Buffered Saline (PBS) placebo (3 mL) and followed up for 13 weeks in previous study (NCT00449696). After completion of previous study, patients entered this study and received 1 single dose of Gel-200 (3mL) intra-articular injection into knee joint.
Period: Overall Study
Arm/Group | 2Gel-200 | 1PBS1Gel-200
Started | 125 | 77
Received Injection | 125 | 74
Analyzed Participants | 122 (3 subjects removed from ITT analyses because of no post treatment data (pre-defined criteria).) | 74
Completed | 112 | 71
Not Completed | 13 | 6
Not completed — Other Treatment Required | 5 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Others | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2Gel-200 | 1PBS1Gel-200 | Total
Number analyzed (Participants) | 122 | 74 | 196
Age Continuous [Mean (Standard Deviation); unit: years] | 61.4 (10.29) | 61.6 (10.50) | 61.4 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 48 | 122
  Male | 48 | 26 | 74
Region of Enrollment [Number; unit: participants]
  United States | 122 | 74 | 196
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/meters square] | 28.6 (4.14) | 29.1 (4.01) | 28.8 (4.09)
WOMAC VAS Pain Subscore [Mean (Standard Deviation); unit: Scores on a scale] — Assessed Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Visual Analog Scale (VAS) pain subscores on VAS of 100 mm.; 0 mm meaning no pain; 100 mm meaning extreme pain.
  Scores on a scale | 69.4 (15.82) | 69.9 (15.13) | 69.5 (15.53)
WOMAC VAS Stiffness Subscore [Mean (Standard Deviation); unit: scores on a scale] — Assessed Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Visual Analog Scale (VAS) stiffness subscores on VAS of 100 mm.; 0 mm meaning no stiffness; 100 mm meaning extreme stiffness.
  scores on a scale | 69.7 (18.31) | 70.7 (18.40) | 70.1 (18.30)
WOMAC VAS Physical Function Subcore [Mean (Standard Deviation); unit: scores on a scale] — Assessed Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Visual Analog Scale (VAS) physical function subscores on VAS of 100 mm.; 0 mm meaning no difficulty; 100 mm meaning extreme difficulty.
  scores on a scale | 68.0 (17.96) | 69.9 (16.35) | 68.7 (17.35)
WOMAC VAS Total Score [Mean (Standard Deviation); unit: scores on a scale] — Mean of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Visual Analog Scale (VAS) pain, stiffness and physical function subscores on VAS of 100 mm.; 0 mm meaning no pain, stiffness and difficulty; 100 mm meaning extreme pain, stiffness and difficulty.
  scores on a scale | 68.4 (17.07) | 69.9 (15.79) | 69.0 (16.58)
Subject Global Evaluations [Mean (Standard Deviation); unit: scores on a scale] — Observed subject evaluations on Visual Analog Scale (VAS) of 100 mm.; 0 mm meaning excellent feeling in knee joint; 100 mm meaning poor feeling in knee joint.
  scores on a scale | 66.1 (21.81) | 68.2 (18.85) | 66.9 (20.70)
Physician Global Evaluations [Mean (Standard Deviation); unit: scores on a scale] — Observed physician evaluations on Visual Analog Scale (VAS) of 100 mm.; 0 mm meaning excellent feeling in knee joint; 100 mm meaning poor feeling in knee joint.
  scores on a scale | 60.5 (16.85) | 62.6 (20.51) | 61.3 (18.29)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Systemic and Local Adverse Events Following a Single or Repeat Intra-articular Injection of Gel-200
Time Frame: 13 weeks
Measure: Number; unit: participants
Arm/Group | 2Gel-200 | 1PBS1Gel-200
Number analyzed (Participants) | 125 | 74
participants | 68 | 43
Statistical Analysis 1: Comparison: 2Gel-200 vs 1PBS1Gel-200; Test type: Superiority or Other; p > 0.1, Fisher Exact

2. Secondary Outcome: Improvement From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Visual Analog Scale (VAS) (Pain Subscore)
Description: Observed WOMAC pain subscore on VAS of 100 mm.; 0 mm meaning no pain; 100 mm meaning extreme pain. Improved score from baseline to week 13 were calculated as baseline minus week 13.
Time Frame: Baseline and Week 13
Population: ITT population was used for analysis. 3 patients with 2Gel-200 were removed from ITT population analysis and baseline because of no post treatment data according to a pre-specified rule. These data were submitted to FDA.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | 2Gel-200 | 1PBS1Gel-200
Number analyzed (Participants) | 122 | 74
millimeters | 32.3 (22.68) | 35.4 (22.97)
Statistical Analysis 1: Comparison: 2Gel-200; One-sample 2 sided t-test of change from baseline within 2Gel-200 group; no between-group test was performed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: 1PBS1Gel-200; One-sample 2 sided t-test of change from baseline within 1PBS1Gel-200 group; no between-group test was performed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Improvement From Baseline in WOMAC VAS (Stiffness Subscore)
Description: Observed WOMAC stiffness subscore on Visual Analog Scale (VAS) of 100 mm; 0 mm meaning no stiffness; 100 mm meaning extreme stiffness. Improved score from baseline to week 13 were calculated as baseline minus week 13.
Time Frame: Baseline and Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | 2Gel-200 | 1PBS1Gel-200
Number analyzed (Participants) | 122 | 74
millimeters | 29.0 (24.95) | 34.5 (25.27)
Statistical Analysis 1: Comparison: 2Gel-200; One-sample 2 sided t-test of change from baseline within 2Gel-200 group; no between-group test was performed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: 1PBS1Gel-200; One-sample 2 sided t-test of change from baseline within 1PBS1Gel-200 group; no between-group test was performed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

4. Secondary Outcome: Improvement From Baseline in WOMAC VAS (Physical Function Subscore)
Description: Observed WOMAC physical function subscore on Visual Analog Scale (VAS) of 100 mm; 0 mm meaning no difficulty; 100 mm meaning extreme difficulty. Improved score from baseline to week 13 were calculated as baseline minus week 13.
Time Frame: Baseline and Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | 2Gel-200 | 1PBS1Gel-200
Number analyzed (Participants) | 122 | 74
millimeters | 30.1 (22.85) | 34.4 (24.04)
Statistical Analysis 1: Comparison: 2Gel-200; One-sample 2 sided t-test of change from baseline within 2Gel-200 group; no between-group test was performed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: 1PBS1Gel-200; One-sample 2 sided t-test of change from baseline within 1PBS1Gel-200 group; no between-group test was performed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

5. Secondary Outcome: Improvement From Baseline in WOMAC VAS (Total Score)
Description: Observed all WOMAC mean scores on Visual Analog Scale (VAS) of 100 mm; a total of WOMAC pain, stiffness, and physical function subscores. Improved score from baseline to week 13 were calculated as baseline minus week 13.
Time Frame: Baseline and Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | 2Gel-200 | 1PBS1Gel-200
Number analyzed (Participants) | 122 | 74
millimeters | 30.4 (22.60) | 34.6 (23.66)
Statistical Analysis 1: Comparison: 2Gel-200; One-sample 2 sided t-test of change from baseline within 2Gel-200 group; no between-group test was performed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: 1PBS1Gel-200; One-sample 2 sided t-test of change from baseline within 1PBS1Gel-200 group; no between-group test was performed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Outcome Measures in Rheumatology Artthritis Clinical Trials (OMERACT) - and the Osteoarthritis Research Society International (OARSI) Response
Description: Outcome Measures in Rheumatology Clinical Trials and Osteoarthritis Research Society International (OMERACT-OARSI) strict responses defined by improvements from baseline in WOMAC pain or physical function subscore ≥50% with absolute changes ≥20 mm (termed strict responders), or ≥20% with absolute changes ≥10mm in 2 of 3 measures of WOMAC pain or physical function subscore or subject global evaluations (termed responders).
Time Frame: Weeks 13
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | 2Gel-200 | 1PBS1Gel-200
Number analyzed (Participants) | 122 | 74
Percentage of Participants
  Participants who met strict responders at week 13 | 58.0 | 57.7
  Participants who met responders at week 13 | 75.0 | 77.5

7. Secondary Outcome: Improvement From Baseline in Subject Global Evaluations
Description: Observed subject evaluations on Visual Analog Scale (VAS) of 100 mm; 0 mm meaning excellent feeling in knee joint; 100 mm meaning poor feeling in knee joint. Improved score from baseline to week 13 were calculated as baseline minus week 13.
Time Frame: Baseline and Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | 2Gel-200 | 1PBS1Gel-200
Number analyzed (Participants) | 122 | 74
millimeters | 29.8 (30.76) | 33.4 (26.24)
Statistical Analysis 1: Comparison: 2Gel-200; One-sample 2 sided t-test of change from baseline within 2Gel-200 group; no between-group test was performed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: 1PBS1Gel-200; One-sample 2 sided t-test of change from baseline within 1PBS1Gel-200 group; no between-group test was performed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

8. Secondary Outcome: Improvement From Baseline in Physician Global Evaluations
Description: Observed physician evaluations on Visual Analog Scale (VAS) of 100 mm; 0 mm meaning excellent feeling in knee joint; 100 mm meaning poor feeling in knee joint. Improved score from baseline to week 13 were calculated as baseline minus week 13.
Time Frame: Baseline and Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | 2Gel-200 | 1PBS1Gel-200
Number analyzed (Participants) | 122 | 74
millimeters | 27.4 (25.08) | 27.4 (27.15)
Statistical Analysis 1: Comparison: 2Gel-200; One-sample 2 sided t-test of change from baseline within 2Gel-200 group; no between-group test was performed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: 1PBS1Gel-200; One-sample 2 sided t-test of change from baseline within 1PBS1Gel-200 group; no between-group test was performed; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

9. Secondary Outcome: Acetaminophen Consumption
Description: Weekly mean acetaminophen consumption between weeks 9 and 13.
Time Frame: Week 9 to Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | 2Gel-200 | 1PBS1Gel-200
Number analyzed (Participants) | 122 | 74
milligrams | 1677.4 (3135.80) | 1822.5 (2768.22)

ADVERSE EVENTS:
Arm/Group | 2Gel-200 | 1PBS1Gel-200
Serious Adverse Events (participants affected / at risk) | 3/125 | 1/74
Other Adverse Events (participants affected / at risk) | 44/125 | 27/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2Gel-200 (N=125) | 1PBS1Gel-200 (N=74)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2Gel-200 (N=125) | 1PBS1Gel-200 (N=74)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (18) | 8 (8)
Joint effusion (Musculoskeletal and connective tissue disorders) | 27 (29) | 19 (24)
Joint swelling (Musculoskeletal and connective tissue disorders) | 25 (28) | 17 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
SKK has the right to review the disclosures. Investigator shall not make any publication of study data, results or similar information without the express of permission of SKK.